CLINICAL TRIAL: NCT00579267
Title: Reliability and Validity of the MINI International Neuropsychiatric Interview for Children and Adolescents (MINI-KID)
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: David V. Sheehan, MD, MBA, University of South Florida College of Medicine
Other Study IDs: MINI-KID Validation Study
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2007-12

CONDITIONS: Major Depression; Mania; Anxiety Disorders; Psychotic Disorder; Alcohol Dependence; Drug Dependence; Eating Disorders; Suicidality; Dysthymia; ADHD; Tourettes Disorder; Conduct Disorder; Oppositional Defiant Disorder; Pervasive Developmental Disorder
Keywords: MINI-KID; structured diagnostic interview; reliability and validity; K-SADS; Sheehan Disability Scale
MeSH Terms: conditions — Depressive Disorder, Major; Mania; Anxiety Disorders; Psychotic Disorders; Alcoholism; Substance-Related Disorders; Feeding and Eating Disorders; Suicidal Ideation; Dysthymic Disorder; Attention Deficit Disorder with Hyperactivity; Tourette Syndrome; Conduct Disorder; Oppositional Defiant Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MINI-KID — Structured Diagnostic Interview for children and adolescent psychiatric disorders.

SUMMARY:
The primary aims of this study are to assess:

1. The inter-rater and test-retest reliability of the MINI-KID
2. The validity of the standard MINI-KID interview in relation to the parent rated pencil/paper version (MINI-KID-P) and th longer clinician rated "Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime Version (K-SADS-PL) and "expert opinion" (when available).

Secondary aims will include evaluating the concordance between: The Children's Global Assessment Scale (a required part of the K-SADS) with the clinician-rated Sheehan Disability Scale (to be administered with the MINI-KID) as a measure of illness severity.

DETAILED DESCRIPTION:
The MINI-KID is a short, structured diagnostic interview used to assess the presence of 24 DSM-IV child and adolescent psychiatric disorders as well as the risk of suicide.

To achieve adequate representation of the major psychiatric disorders and sufficient normal controls, we propose recruiting 230 children and adolescents (ages 6 to 17 years 11 months), comprised of 200 subjects identified as having one or more psychiatric disorders and 30 normal controls in the community. These subjects will be from diverse socioeconomic, racial and ethnic backgrounds. We will assess the inter-rater and test-retest reliability of the MINI-KID and examine its validity with the "gold-standard" diagnostic interview for children and adolescents as well as expert opinion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 6 years and 17 years, 11 months
* All subjects must meet MINI-KID DSM-IV criteria for a least one of the Axis I child psychiatry disorders covered by the MINI-KID.
* Both sexes are included.

Exclusion Criteria:

* Subjects who suffer from mental retardation, significant developmental disorders, congenital abnormalities, delirium, dementia, a language problem, or brain damage will be excluded.
* Subjects with neurological disorders, chronic or life threatening diseases will be excluded.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescents between the ages of 6 and 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2004-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Kappa scores between MINI Kid and K-SADS | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David V. Sheehan, MD, MBA, Principal Investigator — University of South Florida College of Medicine
Locations (1):
- University of South Florida College of Medicine, Department of Psychiatry, Tampa, Florida, United States

REFERENCES:
- [Derived] Sheehan DV, Sheehan KH, Shytle RD, Janavs J, Bannon Y, Rogers JE, Milo KM, Stock SL, Wilkinson B. Reliability and validity of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). J Clin Psychiatry. 2010 Mar;71(3):313-26. doi: 10.4088/JCP.09m05305whi. PMID 20331933